CLINICAL TRIAL: NCT06758999
Title: Validity and Reliability of the Turkish Form of the Outpatient Physical Therapy Improvement in Movement Assessment Log
Brief Title: Validity and Reliability of the Turkish Form of the OPTIMAL
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-011
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Outpatient Treatment
Keywords: reliability; validity; outpatient physical therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
The primary aim of the study was to determine the reliability and validity of the Turkish version of the questionnaire named "The Outpatient Physical Therapy Improvement in Movement Assessment Log". The secondary aim of the study was to measure the physical activity and mobility of outpatients receiving physical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older
2. Receiving outpatient physical therapy
3. Volunteering to participate in the study
4. Knowing how to read and write

Exclusion Criteria:

1. Having a cognitive problem that prevents you from completing the survey independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients to be included in the study will be those who are receiving outpatient treatment at the Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center and who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The Outpatient Physical Therapy Improvement in Movement Assessment Log | 20 weeks

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No